CLINICAL TRIAL: NCT03190187
Title: Spinal Manipulation Effectiveness in Pain, Disability and Range of Motion.
Brief Title: Spinal Manipulation Effectiveness in Spinal Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: DAVID CRUZ DÍAZ (Other)
Responsible Party: Sponsor-Investigator, DAVID CRUZ DÍAZ, Physical Therapy Department Coordinator, University of Jaén
Organization: University of Jaén (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ManipulationUja
Record Dates: First submitted 2017-02-24; First posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-06

CONDITIONS: Low Back Pain; Cervical Pain; Pain
MeSH Terms: conditions — Low Back Pain; Neck Pain; Pain | interventions — Manipulation, Spinal

STUDY DESIGN:
Intervention Model Description: Single blind parallel clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients will be randomly allocated to spinal manipulation group or sham group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal manipulation (Active Comparator): Spinal manipulation to the spine will be applied to participants enrolled in this group.
  Interventions: Other: Spinal Manipulation
- Sham manipulation (Sham Comparator): Sham technique wich mimic the intervention manipulation with less force and different body location will be applied.
  Interventions: Other: Sham manipulation

INTERVENTIONS:
Other: Spinal Manipulation — Spinal manipulation based on orthopaedic manual therapy approach
  Arms: Spinal manipulation
Other: Sham manipulation — Patients will receive simulated spinal manipulation without force application
  Arms: Sham manipulation

SUMMARY:
The aim of the present intervention study is to determine the effectiveness of manipulation techniques.

DETAILED DESCRIPTION:
Spinal manipulation of the spine will be assessed in patients with musculoskeletal disorders to determine the effects of different manual therapy approaches.

ELIGIBILITY:
Inclusion Criteria:

* Currently suffering spinal related pain (neck, thoracic or lumbar).
* Not receiving additional treatment for the treated condition.

Exclusion Criteria:

* Presence of red flags such as tumors or infection.
* Recent surgery.
* Fractures.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 98 (Estimated)
Dates: Start 2018-02-20 (Estimated); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Visual analogical scale | Change from baseline to 4 weeks and 6 months of follow up.
  Pain was measured using a visual analogical scale (VAS). The VAS consists of a 10-cm line, with the left extremity representing (absence of pain) and the right extremity indicating (the worse pain devisable). Participants were asked to indicate in the scale their current level of pain being higher values related with more intense pain

SECONDARY OUTCOMES:
Oswestry Disability Index | Change from baseline to 4 weeks and 6 months of follow up.
  The Oswestry Disability Index is a 10 item questionnaire measuring low back pain related disability. Individual item scores range from 0 to 5. Scores on all items are summed and multiplied by 2 to provide a percentage ranging between 0 to 100 with higher scores indicating greater low back pain related disability.
Range of Motion | Change from baseline to 4 weeks and 6 months of follow up.
  The spinal range of motion will be assessed with a digital inclinometer which indicates the results in angular degrees.

CONTACTS AND LOCATIONS:
Overall Officials: DAVID Curz DIAZ, PhD, Principal Investigator — University of Jaen
Locations (1):
- University of Jaen, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No
There is no intention to share the plan